CLINICAL TRIAL: NCT03165773
Title: Four-hour Glycemic Kinetic Response Following 13C-enriched Oatmeal Breakfast Compared to Hot Corn Grits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1503
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Glycemic and Insulinemic Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oatmeal (Experimental): 87 grams oatmeal
  Interventions: Other: Oatmeal
- Corn grits (Active Comparator): 67 grams corn grits
  Interventions: Other: Corn grits

INTERVENTIONS:
Other: Oatmeal — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence
  Arms: Oatmeal
Other: Corn grits — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence
  Arms: Corn grits

SUMMARY:
The objectives of this study are to assess the 4 hr postprandial kinetics of total and exogenous glucose in response to consumption of oatmeal containing a high percentage of the viscous agent β-glucan, in comparison to a β-glucan free corn cereal that is matched by grams of available carbohydrate.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-45 years of age.
* Subject has a body mass index (BMI) between 18.5 and 29.9 kg/m2, inclusive at screening (visit 1).
* Subject has normal fasting serum glucose (<6.5 mmol/L capillary corresponding to whole blood glucose <5.8 mmol/L) at beginning of each visit.
* Subject has no health conditions that would prevent him from fulfilling the study requirements as judged by the Investigator on the basis of medical history.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria.
* Failure to comply with pre-visit instructions on diet and physical activity.
* Known history of clinically important medical conditions, such as any major trauma or surgical event within 3 months of screening, AIDS, cancer, hepatitis, endocrine (including Type 1 and Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary, or GI disorders.
* Subject using medications or supplements known to influence carbohydrate or lipid metabolism, including, but not limited to adrenergic blocks, diuretics, thiazolidinediones, metformin, statins, and systemic corticosteroids within 4 weeks of the screening visit.
* Subject who cannot or will not comply with the experimental procedures or does not follow GI Labs safety guidelines.
* Subject has a known intolerance, sensitivity or allergy to any ingredients in the study products.
* Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Exogenous glucose 0-4 h | 0-4 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, Principal Investigator — GI Labs
Locations (1):
- Glycemic Index Laboratories, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No